CLINICAL TRIAL: NCT01503723
Title: Biomarkers in Exhaled Breath Condensates in Acute Lung Injury: Early Detection and Outcome Predictors
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201103016RC
Record Dates: First submitted 2012-01-02; First posted 2012-01-04 (Estimated); Last update posted 2012-01-04 (Estimated); Status verified 2011-09

CONDITIONS: Acute Lung Injury
MeSH Terms: conditions — Acute Lung Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Exhaled breath condensate
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with acute lung injury: Patients who are admitted to ICU with the diagnosis of acute hypoxemic respiratory failure
  Interventions: Other: Determined by intended physician

INTERVENTIONS:
Other: Determined by intended physician — We perform a prospective observational study. All the treatment for the patients are determined by intended physicians.

SUMMARY:
Metabolomics, or metabonomics, is a large-scale approach to monitoring as many as possible of the compounds involved in cellular processes in a single assay to derive metabolic profiles. Metabolomics allows for a global assessment of a cellular state within the context of the immediate environment, taking into account genetic regulation, altered kinetic activity of enzymes, and changes in metabolic reactions. Metabolomics may be useful for understanding metabolic imbalances and for diagnosis of human disease. The investigators plan to collect exhaled breath condensate from patients with acute lung injury. Metabolomic analysis in the patients may help us to explore some novel biomarkers for the disease diagnosis and outcome prediction.

DETAILED DESCRIPTION:
Acute lung injury (ALI) and acute respiratory distress syndrome (ARDS) are the leading causes of mortality and morbidity in the intensive care unit (ICU). The causes of ALI/ARDS differ from patient to patient, including sepsis, aspiration, systemic inflammation, trauma, blood transfusion, etc. With early detection and treatment, the survival rate may be improved significantly. However, it is often difficult to differentiate ALI/ARDS from cardiogenic pulmonary edema or other causes, even with advanced technology and invasive tools. A potential tool is the breath chemical test, ranging from exhaled gas measurement, such as exhaled nitric oxide or carbonic monoxide, to volatile organic compound determination and nonvolatile biomarker profiling. Being completely noninvasive, sampling of the exhaled breath condensates (EBC) allows clinicians and researchers to assess body functions in an easier and flexible manner. Exhaled breath contains thousands of volatile and nonvolatile compounds in trace amounts. Therefore, it is not until recently, after the development of highly sensitive cutting-edge technologies in sample analysis, that the evaluation of this type of human specimens becomes possible. Advanced technologies in proteomics, metabolomics, GC/LC-Mass Spectrometry and pattern recognition computation generate a field of exhaled biomarker profiling, called "breathomics." After the establishment of the metabolomic profiling of EBC in patients with ALI, ARDS or cardiogenic pulmonary edema, a useful and powerful noninvasive tool for ALI/ARDS diagnosis and outcome prediction could be set up.

Metabolomics, or metabonomics, is a large-scale approach to monitoring as many as possible of the compounds involved in cellular processes in a single assay to derive metabolic profiles. Although metabolomics first referred to the monitoring of individual cells and metabonomics referred to multicellular organisms, these terms are now often used interchangeably. Metabolic changes occur through a number of mechanisms, including direct genetic regulation and alterations in enzymatic and metabolic reactions. Metabolomics allows for a global assessment of a cellular state within the context of the immediate environment, taking into account genetic regulation, altered kinetic activity of enzymes, and changes in metabolic reactions. Thus, compared with genomics or proteomics, metabolomics reflects changes in phenotype and therefore function. Techniques applied to metabolic profiling include nuclear magnetic resonance (NMR) and mass spectrometry (MS). Metabolomics have the advantage of being capable of searching for proteins or metabolites in the blood or urine. Metabolomics may be useful for understanding metabolic imbalances and for diagnosis of human disease. Over 30 endogenous metabolites have been studied in breast tissue, and breast cancer show elevated total choline-containing compounds (tCho), low glycerophosphocholine, and low glucose compared with benign tumors or healthy tissue. Similar to breast cancer, prostate cancer exhibits a distinct metabolic profile characterized by high tCho and phosphocholine levels, along with an increase in the glycolytic products lactate and alanine. In prostate cancer, citrate may also be a marker of responsiveness to treatment. These results show the potential utility of metabolomics in cancer diagnosis and clinical evaluation.

Breath chemical tests have a broad spectrum of applications ranging from exhaled nitric oxide fraction (FeNO) measurement to monitor the effect of anti-inflammatory treatment in asthma, to volatile organic compound (VOC) determination and nonvolatile biomarker profiling in the cooled breath sample called exhaled breath condensate (EBC). Being completely noninvasive, sampling of the breath allows clinicians and researchers to assess different body functions in a flexible manner. Therefore, breath testing is considered to be a potentially ideal candidate for screening purposes. Besides widely known constituents such as nitrogen, oxygen, carbon dioxide, inert gases and water vapour, exhaled breath also consists of thousands of volatile and nonvolatile components, mainly in trace amounts, making detection a challenging task. The use of innovative "-omics" technologies, including proteomics, metabolomics, mass spectromics, gas chromatography/mass spectrometry (GC-MS) and ion mobility spectrometries, offers great potential for the field of exhaled biomarker profiling. Unlike bronchoalveolar lavage (BAL) and sputum induction which involves inhalation of hypertonic saline to induce cough and possibly bronchoconstriction, EBC does not influence airway function or cause inflammation. It can be easily and safely performed on patients with severe illness and even allows for repeated measurements to be taken. As such, this is a relatively new field with potential for more studies to be performed to investigate acute lung injury by metabolomics.

ELIGIBILITY:
Inclusion Criteria:

* above 18 years old
* admitted to ICU with the diagnosis of acute hypoxemic respiratory failure and endotracheally intubated with mechanical ventilation.

Exclusion Criteria:

* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are admitted to ICU with the diagnosis of acute hypoxemic respiratory failure and endotracheally intubated with mechanical ventilation.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2011-08

PRIMARY OUTCOMES:
Diagnosis | 28 days
  To differentiate ALI/ARDS from cardiogenic pulmonary edema or other causes
Disease severity | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Lu-Cheng Kuo, MD, Master, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan